CLINICAL TRIAL: NCT03510117
Title: Creating and Optimizing Mindfulness Measures to Enhance and Normalize Clinical Evaluation (COMMENCE)
Brief Title: Creating and Optimizing Mindfulness Measures to Enhance and Normalize Clinical Evaluation
Acronym: COMMENCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University of Pittsburgh (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, David Victorson, Associate Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STU00205373; 1R01AT009539-01 (NIH)
Record Dates: First submitted 2018-04-16; First posted 2018-04-27 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Mindfulness
Keywords: Mindfulness; Patient reported outcomes measures; PROMIS
MeSH Terms: interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: To evaluate different forms of validity (e.g., construct, criterion), responsiveness to change over time, and estimation of minimally important differences, we will administer new mindfulness short forms, legacy measures, and an experiential measure of focused attention to ~250 mindfulness students at baseline, 8-weeks, and 16 weeks in multiple, on-going 8-week Mindfulness-Based Stress Reduction (MBSR) courses and similar MBI programs at Pittsburgh and Chicago sites, as well as at member sites from the Academic Consortium for Integrative Medicine and Health and the BraveNet Practice-Based Research Network.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness (Other): Mindfulness
  Interventions: Behavioral: Mindfulness

INTERVENTIONS:
Behavioral: Mindfulness — Mindfulness

SUMMARY:
While MBI trials have reached a greater level of rigor (e.g., random assignment, matching on time, attention, teacher characteristics, non-specific factors) a significant gap still remains in mindfulness research: the lack of a comprehensive and standardized self-report measurement system. A precise, carefully constructed set of assessment tools based on a common measurement system are needed; where scores can be psychometrically linked to current "legacy" measures to better understand the existing body of mindfulness research. In this study, Creating and Optimizing Mindfulness Measures to Enhance and Normalize Clinical Evaluation (COMMENCE), the investigators will use Patient Reported Outcomes Measurement Information System (PROMIS) methodologies to construct improved self-report mindfulness-related measures. They will also use PROMIS-based PROsetta Stone linking methods to equate scores and create cross-walks between new mindfulness measures and existing ones.

DETAILED DESCRIPTION:
The investigators will use Patient Reported Outcomes Measurement Information System (PROMIS®) methodologies to construct improved self-report mindfulness-related measures. They will also use PROMIS-based PROsetta Stone® instrument linking methods to equate scores and create cross-walks between new mindfulness measures and existing ones. The research team has extensive experience in patient reported outcomes (PRO) development through PROMIS and related PRO development initiatives, including mind-body measures (Chicago and Pittsburgh), PROsetta Stone linking methodologies (Chicago), and mindfulness research (Pittsburgh and Chicago).

PROMIS methodologies involve a systematic and iterative approach to person-centered measurement and are the gold standard. Following PROMIS methods, newly created mindfulness measures will be informed by: 1) the existing literature, and 2) stakeholders such as mindfulness researchers, Buddhist and MBI teachers, and new and experienced meditators. COMMENCE analyses will also reflect PROMIS, producing concise, precise, clinically relevant measures that can be administered as Computerized Adaptive Tests (CATs) or fixed-length short forms. PROsetta Stone methods will enable a crosswalk between the new mindfulness measures and legacy instruments that assess similar constructs. All of this will have a major impact on mindfulness research through increasing measurement precision and comparability across and between studies: past, present, and future. The project will also address the response shift challenge. New mindfulness measures and crosswalk linking will be produced through the following three SPECIFIC AIMS:

SPECIFIC AIM I. Development of New Mindfulness Item Banks. Activities include: 1) a review of the mindfulness measurement literature; 2) an online survey of mindfulness researchers to identify domains and measurement considerations for item bank development; 3) focus groups with new and experienced meditators, and individual interviews with mindfulness meditation practitioners, including Buddhist teachers, to elaborate on concepts such as response shift; 4) item refinement; 6) translatability review; and 7) cognitive interviews to assess item clarity.

SPECIFIC AIM II. Calibration of New Mindfulness Item Banks and Score Linking with Legacy Measures. Calibration activities will include: 1) testing new mindfulness item banks in a large online general population sample (n=4200) and a sample of mindfulness teachers and students (n=500); 2) evaluation of dimensionality and other assumptions prior to Item Response Theory (IRT) analysis; 3) IRT analyses; and 4) creation of CATs and fixed length short forms. A battery of legacy measures will also be administrated alongside new mindfulness banks. Using PROsetta Stone procedures, the investigators will test mindfulness banks and legacy measures in a new large online sample (n=3000) to link measures on a common measurement metric and create cross-walk scoring tables to facilitate interpretation.

SPECIFIC AIM III. Validation of New Mindfulness Short Forms in Ongoing Mindfulness Courses. To evaluate different forms of validity (e.g., construct, criterion), responsiveness to change over time, and estimation of minimally important differences, the investigators will administer new mindfulness short forms and legacy measures to 250 mindfulness students at baseline, 8-weeks, and 16 weeks in multiple, on-going 8-week Mindfulness-Based Stress Reduction (MBSR) courses and similar MBI programs at Pittsburgh and Chicago sites, as well as at member sites from the Academic Consortium for Integrative Medicine and Health and the BraveNet Practice-Based Research Network. In addition to legacy measures, a subset of the sample will complete the meditation breath awareness score, an experiential measure of focused attention.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years of age
* Must be able to speak and understand English
* Must be enrolled in an multi-week, group-based, instructor-led, live (in-person or online) mindfulness-based program that has not yet started (i.e., before session 1)

Exclusion Criteria:

* Unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8152 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2022-07-26 (Actual); Study Completion 2022-07-26 (Actual)

PRIMARY OUTCOMES:
Mindfulness Questionnaire | DAY 0
  Mindfulness Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: David E Victorson, PhD, Principal Investigator — Northwestern University
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chuang tsu: Basic writings. B. Watson, Trans. ed. New York: Columbia University Press; 1964
- [Background] Kabat-Zinn J. Full catastrophe living : using the wisdom of your body and mind to face stress, pain, and illness. Revised and updated edition. ed. New York: Bantam Books trade paperback; 2013
- [Background] Teasdale JD, Segal Z, Williams JM. How does cognitive therapy prevent depressive relapse and why should attentional control (mindfulness) training help? Behav Res Ther. 1995 Jan;33(1):25-39. doi: 10.1016/0005-7967(94)e0011-7. PMID 7872934
- [Background] Linehan MM. Dialectical behavior therapy for borderline personality disorder. Theory and method. Bull Menninger Clin. 1987 May;51(3):261-76. No abstract available. PMID 3580661
- [Background] Hayes SC, Wilson KG. Acceptance and commitment therapy: Altering the verbal support for experiential avoidance. Behav Anal. 1994 Fall;17(2):289-303. doi: 10.1007/BF03392677. PMID 22478193
- [Background] Veehof MM, Trompetter HR, Bohlmeijer ET, Schreurs KM. Acceptance- and mindfulness-based interventions for the treatment of chronic pain: a meta-analytic review. Cogn Behav Ther. 2016;45(1):5-31. doi: 10.1080/16506073.2015.1098724. Epub 2016 Jan 28. PMID 26818413
- [Background] Morone NE, Greco CM, Moore CG, Rollman BL, Lane B, Morrow LA, Glynn NW, Weiner DK. A Mind-Body Program for Older Adults With Chronic Low Back Pain: A Randomized Clinical Trial. JAMA Intern Med. 2016 Mar;176(3):329-37. doi: 10.1001/jamainternmed.2015.8033. PMID 26903081
- [Background] Grossman P, Zwahlen D, Halter JP, Passweg JR, Steiner C, Kiss A. A mindfulness-based program for improving quality of life among hematopoietic stem cell transplantation survivors: feasibility and preliminary findings. Support Care Cancer. 2015 Apr;23(4):1105-12. doi: 10.1007/s00520-014-2452-4. Epub 2014 Oct 10. PMID 25297466
- [Background] Victorson D, Hankin V, Burns J, Weiland R, Maletich C, Sufrin N, Schuette S, Gutierrez B, Brendler C. Feasibility, acceptability and preliminary psychological benefits of mindfulness meditation training in a sample of men diagnosed with prostate cancer on active surveillance: results from a randomized controlled pilot trial. Psychooncology. 2017 Aug;26(8):1155-1163. doi: 10.1002/pon.4135. Epub 2016 May 3. PMID 27145355
- [Background] Slowikowski C, Mioduszewski O, MacLean H, Poulin P, Smith AM, Walker LAS. Mindfulness, mood and quality of life in multiple sclerosis. Mult Scler J. 2016;22:47-47
- [Background] Eisendrath SJ, Gillung E, Delucchi KL, Segal ZV, Nelson JC, McInnes LA, Mathalon DH, Feldman MD. A Randomized Controlled Trial of Mindfulness-Based Cognitive Therapy for Treatment-Resistant Depression. Psychother Psychosom. 2016;85(2):99-110. doi: 10.1159/000442260. Epub 2016 Jan 26. PMID 26808973
- [Background] Maxwell L, Duff E. Mindfulness: An Effective Prescription for Depression and Anxiety. Jnp-J Nurse Pract. 2016;12(6):403-409
- [Background] Brown KW, Weinstein N, Creswell JD. Trait mindfulness modulates neuroendocrine and affective responses to social evaluative threat. Psychoneuroendocrinology. 2012 Dec;37(12):2037-41. doi: 10.1016/j.psyneuen.2012.04.003. Epub 2012 May 22. PMID 22626868
- [Background] Creswell JD, Pacilio LE, Lindsay EK, Brown KW. Brief mindfulness meditation training alters psychological and neuroendocrine responses to social evaluative stress. Psychoneuroendocrinology. 2014 Jun;44:1-12. doi: 10.1016/j.psyneuen.2014.02.007. Epub 2014 Feb 23. PMID 24767614
- [Background] Creswell JD, Irwin MR, Burklund LJ, Lieberman MD, Arevalo JM, Ma J, Breen EC, Cole SW. Mindfulness-Based Stress Reduction training reduces loneliness and pro-inflammatory gene expression in older adults: a small randomized controlled trial. Brain Behav Immun. 2012 Oct;26(7):1095-101. doi: 10.1016/j.bbi.2012.07.006. Epub 2012 Jul 20. PMID 22820409
- [Background] Creswell JD, Taren AA, Lindsay EK, Greco CM, Gianaros PJ, Fairgrieve A, Marsland AL, Brown KW, Way BM, Rosen RK, Ferris JL. Alterations in Resting-State Functional Connectivity Link Mindfulness Meditation With Reduced Interleukin-6: A Randomized Controlled Trial. Biol Psychiatry. 2016 Jul 1;80(1):53-61. doi: 10.1016/j.biopsych.2016.01.008. Epub 2016 Jan 29. PMID 27021514
- [Background] Davidson RJ, Kabat-Zinn J, Schumacher J, Rosenkranz M, Muller D, Santorelli SF, Urbanowski F, Harrington A, Bonus K, Sheridan JF. Alterations in brain and immune function produced by mindfulness meditation. Psychosom Med. 2003 Jul-Aug;65(4):564-70. doi: 10.1097/01.psy.0000077505.67574.e3. PMID 12883106
- [Background] Ferrarelli F, Smith R, Dentico D, Riedner BA, Zennig C, Benca RM, Lutz A, Davidson RJ, Tononi G. Experienced mindfulness meditators exhibit higher parietal-occipital EEG gamma activity during NREM sleep. PLoS One. 2013 Aug 28;8(8):e73417. doi: 10.1371/journal.pone.0073417. eCollection 2013. PMID 24015304
- [Background] Cullen M. Mindfulness-Based Interventions: An Emerging Phenomenon. Mindfulness. 2011;2:186-193
- [Background] Kabat-Zinn J. Full Catastrophe Living: Using the Wisdom of your Mind to Face Stress, Pain and Illness. New York: Dell Publishing; 1990
- [Background] Quaglia JT, Braun SE, Freeman SP, McDaniel MA, Brown KW. Meta-analytic evidence for effects of mindfulness training on dimensions of self-reported dispositional mindfulness. Psychol Assess. 2016 Jul;28(7):803-18. doi: 10.1037/pas0000268. Epub 2016 Apr 14. PMID 27078183
- [Background] Grossman P. Defining mindfulness by how poorly I think I pay attention during everyday awareness and other intractable problems for psychology's (re)invention of mindfulness: comment on Brown et al. (2011). Psychol Assess. 2011 Dec;23(4):1034-40; discussion 1041-6. doi: 10.1037/a0022713. PMID 22122674
- [Background] Walach H, Buchheld N, Buttenmuller V, Kleinknecht N, Schmidt S. Measuring mindfulness - the Freiburg Mindfulness Inventory (FMI). Personality and Individual Differences. 2006;40(8):1543-1555
- [Background] Baer RA, Smith GT, Allen KB. Assessment of mindfulness by self-report: the Kentucky inventory of mindfulness skills. Assessment. 2004 Sep;11(3):191-206. doi: 10.1177/1073191104268029. PMID 15358875
- [Background] Van Dam NT, Earleywine M, Borders A. Measuring mindfulness? An Item Response Theory analysis of the Mindful Attention Awareness Scale. Personality and Individual Differences. 2010;49(7):805-810
- [Background] Baer RA, Smith GT, Lykins E, Button D, Krietemeyer J, Sauer S, Walsh E, Duggan D, Williams JM. Construct validity of the five facet mindfulness questionnaire in meditating and nonmeditating samples. Assessment. 2008 Sep;15(3):329-42. doi: 10.1177/1073191107313003. Epub 2008 Feb 29. PMID 18310597
- [Background] Schwartz CE, Sprangers MA. Methodological approaches for assessing response shift in longitudinal health-related quality-of-life research. Soc Sci Med. 1999 Jun;48(11):1531-48. doi: 10.1016/s0277-9536(99)00047-7. PMID 10400255
- [Background] Sprangers MA, Schwartz CE. Integrating response shift into health-related quality of life research: a theoretical model. Soc Sci Med. 1999 Jun;48(11):1507-15. doi: 10.1016/s0277-9536(99)00045-3. PMID 10400253
- [Background] Davidson RJ. Empirical explorations of mindfulness: conceptual and methodological conundrums. Emotion. 2010 Feb;10(1):8-11. doi: 10.1037/a0018480. PMID 20141297
- [Background] Morone NE, Rollman BL, Moore CG, Li Q, Weiner DK. A mind-body program for older adults with chronic low back pain: results of a pilot study. Pain Med. 2009 Nov;10(8):1395-407. doi: 10.1111/j.1526-4637.2009.00746.x. PMID 20021599
- [Background] Cherkin DC, Sherman KJ, Turner JA. Mindfulness-Based Stress Reduction vs Cognitive Behavioral Therapy for Chronic Low Back Pain--Reply. JAMA. 2016 Aug 9;316(6):663-4. doi: 10.1001/jama.2016.7951. No abstract available. PMID 27532924
- [Background] Park T, Reilly-Spong M, Gross CR. Mindfulness: a systematic review of instruments to measure an emergent patient-reported outcome (PRO). Qual Life Res. 2013 Dec;22(10):2639-59. doi: 10.1007/s11136-013-0395-8. Epub 2013 Mar 29. PMID 23539467
- [Background] Cella D, Riley W, Stone A, Rothrock N, Reeve B, Yount S, Amtmann D, Bode R, Buysse D, Choi S, Cook K, Devellis R, DeWalt D, Fries JF, Gershon R, Hahn EA, Lai JS, Pilkonis P, Revicki D, Rose M, Weinfurt K, Hays R; PROMIS Cooperative Group. The Patient-Reported Outcomes Measurement Information System (PROMIS) developed and tested its first wave of adult self-reported health outcome item banks: 2005-2008. J Clin Epidemiol. 2010 Nov;63(11):1179-94. doi: 10.1016/j.jclinepi.2010.04.011. Epub 2010 Aug 4. PMID 20685078
- [Background] Pilkonis PA, Yu L, Dodds NE, Johnston KL, Lawrence SM, Daley DC. Validation of the alcohol use item banks from the Patient-Reported Outcomes Measurement Information System (PROMIS). Drug Alcohol Depend. 2016 Apr 1;161:316-22. doi: 10.1016/j.drugalcdep.2016.02.014. Epub 2016 Feb 17. PMID 26936412
- [Background] Sung VW, Griffith JW, Rogers RG, Raker CA, Clark MA. Item bank development, calibration and validation for patient-reported outcomes in female urinary incontinence. Qual Life Res. 2016 Jul;25(7):1645-54. doi: 10.1007/s11136-015-1222-1. Epub 2016 Jan 6. PMID 26732514
- [Background] Dampier C, Jaeger B, Gross HE, Barry V, Edwards L, Lui Y, DeWalt DA, Reeve BB. Responsiveness of PROMIS(R) Pediatric Measures to Hospitalizations for Sickle Pain and Subsequent Recovery. Pediatr Blood Cancer. 2016 Jun;63(6):1038-45. doi: 10.1002/pbc.25931. Epub 2016 Feb 8. PMID 26853841
- [Background] Howell CR, Gross HE, Reeve BB, DeWalt DA, Huang IC. Known-groups validity of the Patient-Reported Outcomes Measurement Information System (PROMIS((R))) in adolescents and young adults with special healthcare needs. Qual Life Res. 2016 Jul;25(7):1815-23. doi: 10.1007/s11136-016-1237-2. Epub 2016 Feb 12. PMID 26872912
- [Background] Greco CM, Glick RM, Morone NE, Schneider MJ. Addressing the "It Is Just Placebo" Pitfall in CAM: Methodology of a Project to Develop Patient-Reported Measures of Nonspecific Factors in Healing. Evid Based Complement Alternat Med. 2013;2013:613797. doi: 10.1155/2013/613797. Epub 2013 Dec 19. PMID 24454501
- [Background] Greco CM, Yu L, Johnston KL, Dodds NE, Morone NE, Glick RM, Schneider MJ, Klem ML, McFarland CE, Lawrence S, Colditz J, Maihoefer CC, Jonas WB, Ryan ND, Pilkonis PA. Measuring nonspecific factors in treatment: item banks that assess the healthcare experience and attitudes from the patient's perspective. Qual Life Res. 2016 Jul;25(7):1625-34. doi: 10.1007/s11136-015-1178-1. Epub 2015 Nov 12. PMID 26563249
- [Background] Victorson D, Tulsky DS, Kisala PA, Kalpakjian CZ, Weiland B, Choi SW. Measuring resilience after spinal cord injury: Development, validation and psychometric characteristics of the SCI-QOL Resilience item bank and short form. J Spinal Cord Med. 2015 May;38(3):366-76. doi: 10.1179/2045772315Y.0000000016. PMID 26010971
- [Background] Victorson DE, Choi S, Judson MA, Cella D. Development and testing of item response theory-based item banks and short forms for eye, skin and lung problems in sarcoidosis. Qual Life Res. 2014 May;23(4):1301-13. doi: 10.1007/s11136-013-0567-6. Epub 2013 Nov 9. PMID 24214179
- [Background] Victorson D, Beaumont JL, Mahadevan R, Grimone A, Burns V, Murry W, Gutierrez S, Schuette S, Brady C, Ring M. Acupuncture-Related Quality of Life Changes Using PROMIS Computer Adaptive Tests in a Pragmatic Trial with Oncology and General Integrative Medicine Patients: The Role of Baseline Acupuncture Expectations. J Altern Complement Med. 2016 Oct;22(10):778-787. doi: 10.1089/acm.2015.0121. Epub 2016 Jul 28. PMID 27467506
- [Background] Schalet BD, Rothrock NE, Hays RD, Kazis LE, Cook KF, Rutsohn JP, Cella D. Linking Physical and Mental Health Summary Scores from the Veterans RAND 12-Item Health Survey (VR-12) to the PROMIS((R)) Global Health Scale. J Gen Intern Med. 2015 Oct;30(10):1524-30. doi: 10.1007/s11606-015-3453-9. Epub 2015 Jul 16. PMID 26179820
- [Background] Schalet BD, Revicki DA, Cook KF, Krishnan E, Fries JF, Cella D. Establishing a Common Metric for Physical Function: Linking the HAQ-DI and SF-36 PF Subscale to PROMIS((R)) Physical Function. J Gen Intern Med. 2015 Oct;30(10):1517-23. doi: 10.1007/s11606-015-3360-0. PMID 25990189
- [Background] Zeng X, Wei J, Oei TP, Liu X. The Self-Compassion Scale is Not Validated in a Buddhist Sample. J Relig Health. 2016 Dec;55(6):1996-2009. doi: 10.1007/s10943-016-0205-z. PMID 26979311
- [Background] Sharf RH. Is mindfulness Buddhist? (and why it matters). Transcult Psychiatry. 2015 Aug;52(4):470-84. doi: 10.1177/1363461514557561. Epub 2014 Oct 31. PMID 25361692
- [Background] Frewen P, Hargraves H, DePierro J, D'Andrea W, Flodrowski L. Meditation Breath Attention Scores (MBAS): Development and investigation of an internet-based assessment of focused attention during meditation practice. Psychol Assess. 2016 Jul;28(7):830-40. doi: 10.1037/pas0000283. Epub 2016 Apr 14. PMID 27078182
- [Background] Frewen PA, Unholzer F, Logie-Hagan KRJ, MacKinley JD. Meditation Breath Attention Scores (MBAS): Test-Retest Reliability and Sensitivity to Repeated Practice. Mindfulness. 2014;5(2):161-169
- [Background] Pilkonis PA, Yu L, Colditz J, Dodds N, Johnston KL, Maihoefer C, Stover AM, Daley DC, McCarty D. Item banks for alcohol use from the Patient-Reported Outcomes Measurement Information System (PROMIS): use, consequences, and expectancies. Drug Alcohol Depend. 2013 Jun 1;130(1-3):167-77. doi: 10.1016/j.drugalcdep.2012.11.002. Epub 2012 Dec 1. PMID 23206377
- [Background] Pilkonis PA, Yu L, Dodds NE, Johnston KL, Maihoefer CC, Lawrence SM. Validation of the depression item bank from the Patient-Reported Outcomes Measurement Information System (PROMIS) in a three-month observational study. J Psychiatr Res. 2014 Sep;56:112-9. doi: 10.1016/j.jpsychires.2014.05.010. Epub 2014 May 29. PMID 24931848
- [Background] Yu L, Buysse DJ, Germain A, Moul DE, Stover A, Dodds NE, Johnston KL, Pilkonis PA. Development of short forms from the PROMIS sleep disturbance and Sleep-Related Impairment item banks. Behav Sleep Med. 2011 Dec 28;10(1):6-24. doi: 10.1080/15402002.2012.636266. PMID 22250775
- [Background] Klem M, Saghafi E, Abromitis R, Stover A, Dew MA, Pilkonis P. Building PROMIS item banks: librarians as co-investigators. Qual Life Res. 2009 Sep;18(7):881-8. doi: 10.1007/s11136-009-9498-7. Epub 2009 Jun 23. PMID 19548118
- [Background] Morone N, Kamprath S, Glick R. Physiologic Measures of Mindfulness Meditation in Older Adults. Journal of General Internal Medicine. 2013;28:S148-S148
- [Background] Morone N, Lynch C, Losasso V, Liebe K, Greco C. Mindfulness to Reduce Psychosocial Stress. Journal of General Internal Medicine. 2011;26:S266-S267
- [Background] Morone NE. Mindfulness helps in chronic pain. Forschende Komplementarmedizin. 2008;15(2):106-108
- [Background] Morone NE, Greco CM. Adapting Mindfulness Meditation for the Older Adult. Mindfulness. 2014;5(5):610-612
- [Background] Morone NE, Greco CM, Weiner DK. Mindfulness meditation for the treatment of chronic low back pain in older adults: a randomized controlled pilot study. Pain. 2008 Feb;134(3):310-319. doi: 10.1016/j.pain.2007.04.038. Epub 2007 Jun 1. PMID 17544212
- [Background] Hankin VV, D.; Polster, R. . Maximizing Acceptance and Enrollment in MBSR Randomized Controlled Trials with Older Men Diagnosed with Cancer. . Poster presented to the 8th Annual International Scientific Conference of Mindfulness in Medicine, Health Care, and Society. Worcester, MA. 2010
- [Background] Victorson D, Du H, Hankin V, et al. MINDFULNESS BASED STRESS REDUCTION DECREASES FEAR OF PROGRESSION OVER TIME FOR MEN WITH PROSTATE CANCER ON ACTIVE SURVEILLANCE: RESULTS FROM A RANDOMIZED CLINICAL TRIAL. The Journal of Urology. 2012;187(4S):384
- [Background] Victorson D, Maletich, C, Gutierrez, B, Schuette, S, Morgan, T, Kutikov, A, Kundu, S, Eggener, S, Brendler, C. Description of a New National Cancer Institute Funded Randomized Controlled Trial
- [Background] Victorson DK, M.; Maletich, C.; Lawton, R.C.; Hankin Kaufman, V.; Borrero, M.; Languido, L.; Lewett, K.; Pancoe, H.; Berkowitz, C. . A Systematic Review and Meta-Analysis of Mindfulness-Based Randomized Controlled Trials Relevant to Lifestyle Medicine. . American Journal of Lifestyle Medicine. 2015;9(3):185-211
- [Background] Epel E, Daubenmier J, Moskowitz JT, Folkman S, Blackburn E. Can meditation slow rate of cellular aging? Cognitive stress, mindfulness, and telomeres. Ann N Y Acad Sci. 2009 Aug;1172:34-53. doi: 10.1111/j.1749-6632.2009.04414.x. PMID 19735238
- [Background] Branstrom R, Kvillemo P, Brandberg Y, Moskowitz JT. Self-report mindfulness as a mediator of psychological well-being in a stress reduction intervention for cancer patients--a randomized study. Ann Behav Med. 2010 May;39(2):151-61. doi: 10.1007/s12160-010-9168-6. PMID 20177843
- [Background] Branstrom R, Duncan LG, Moskowitz JT. The association between dispositional mindfulness, psychological well-being, and perceived health in a Swedish population-based sample. Br J Health Psychol. 2011 May;16(Pt 2):300-16. doi: 10.1348/135910710X501683. Epub 2011 Mar 8. PMID 21489058
- [Background] Duncan LG, Moskowitz JT, Neilands TB, Dilworth SE, Hecht FM, Johnson MO. Mindfulness-based stress reduction for HIV treatment side effects: a randomized, wait-list controlled trial. J Pain Symptom Manage. 2012 Feb;43(2):161-71. doi: 10.1016/j.jpainsymman.2011.04.007. Epub 2011 Sep 17. PMID 21925831
- [Background] Ong JC, Shapiro SL, Manber R. Combining mindfulness meditation with cognitive-behavior therapy for insomnia: a treatment-development study. Behav Ther. 2008 Jun;39(2):171-82. doi: 10.1016/j.beth.2007.07.002. Epub 2007 Nov 14. PMID 18502250
- [Background] Ong JC, Ulmer CS, Manber R. Improving sleep with mindfulness and acceptance: a metacognitive model of insomnia. Behav Res Ther. 2012 Nov;50(11):651-60. doi: 10.1016/j.brat.2012.08.001. Epub 2012 Aug 20. PMID 22975073
- [Background] Perez L, Huang J, Jansky L, Nowinski C, Victorson D, Peterman A, Cella D. Using focus groups to inform the Neuro-QOL measurement tool: exploring patient-centered, health-related quality of life concepts across neurological conditions. J Neurosci Nurs. 2007 Dec;39(6):342-53. doi: 10.1097/01376517-200712000-00005. PMID 18186419
- [Background] Lynch EB, Butt Z, Heinemann A, Victorson D, Nowinski CJ, Perez L, Cella D. A qualitative study of quality of life after stroke: the importance of social relationships. J Rehabil Med. 2008 Jul;40(7):518-23. doi: 10.2340/16501977-0203. PMID 18758667
- [Background] Victorson DE, Cella D, Grund H, Judson MA. A conceptual model of health-related quality of life in sarcoidosis. Qual Life Res. 2014 Feb;23(1):89-101. doi: 10.1007/s11136-013-0438-1. Epub 2013 May 26. PMID 23709098
- [Background] Salsman JM, Victorson D, Choi SW, Peterman AH, Heinemann AW, Nowinski C, Cella D. Development and validation of the positive affect and well-being scale for the neurology quality of life (Neuro-QOL) measurement system. Qual Life Res. 2013 Nov;22(9):2569-80. doi: 10.1007/s11136-013-0382-0. Epub 2013 Mar 23. PMID 23526093
- [Background] Schalet BD, Cook KF, Choi SW, Cella D. Establishing a common metric for self-reported anxiety: linking the MASQ, PANAS, and GAD-7 to PROMIS Anxiety. J Anxiety Disord. 2014 Jan;28(1):88-96. doi: 10.1016/j.janxdis.2013.11.006. Epub 2013 Dec 1. PMID 24508596
- [Background] Castel LD, Williams KA, Bosworth HB, Eisen SV, Hahn EA, Irwin DE, Kelly MA, Morse J, Stover A, DeWalt DA, DeVellis RF. Content validity in the PROMIS social-health domain: a qualitative analysis of focus-group data. Qual Life Res. 2008 Jun;17(5):737-49. doi: 10.1007/s11136-008-9352-3. Epub 2008 May 14. PMID 18478368
- [Background] Victorson D, Manly J, Wallner-Allen K, Fox N, Purnell C, Hendrie H, Havlik R, Harniss M, Magasi S, Correia H, Gershon R. Using the NIH Toolbox in special populations: considerations for assessment of pediatric, geriatric, culturally diverse, non-English-speaking, and disabled individuals. Neurology. 2013 Mar 12;80(11 Suppl 3):S13-9. doi: 10.1212/WNL.0b013e3182872e26. PMID 23479537
- [Background] Zemke R, Kramlinger T. Figuring it Out. Reading, MA: Addison Wesley; 1985
- [Background] Halkitis PN. CAT with a limited item bank. Rasch Measurement Transactions. 1996;9(4):471
- [Background] Lai JS, Cella D, Chang CH, Bode RK, Heinemann AW. Item banking to improve, shorten and computerize self-reported fatigue: an illustration of steps to create a core item bank from the FACIT-Fatigue Scale. Qual Life Res. 2003 Aug;12(5):485-501. doi: 10.1023/a:1025014509626. PMID 13677494
- [Background] Lai JS, Dineen K, Reeve BB, Von Roenn J, Shervin D, McGuire M, Bode RK, Paice J, Cella D. An item response theory-based pain item bank can enhance measurement precision. J Pain Symptom Manage. 2005 Sep;30(3):278-88. doi: 10.1016/j.jpainsymman.2005.03.009. PMID 16183012
- [Background] Schulz EM. Construct deficiency? Rasch Measurement Transactions. 1995;9(3):447
- [Background] Willis GB. Cognitive interviewing: A tool for improving questionnaire design. Thousand Oaks, CA: Sage Publications; 2005
- [Background] Eremenco S, Chang CH, Lent L, Odom L, Ribaudo J, Cella D. Facit multilingual translation project: Version 4 linguistic validation. Quality of Life Research. 1999;8(7):626
- [Background] Chadwick P, Hember M, Symes J, Peters E, Kuipers E, Dagnan D. Responding mindfully to unpleasant thoughts and images: reliability and validity of the Southampton mindfulness questionnaire (SMQ). Br J Clin Psychol. 2008 Nov;47(Pt 4):451-5. doi: 10.1348/014466508X314891. Epub 2008 Jun 20. PMID 18573227
- [Background] Feldman G, Hayes A, Kumar S, Greeson J, Laurenceau JP. Mindfulness and emotion regulation: The development and initial validation of the Cognitive and Affective Mindfulness Scale-Revised (CAMS-R). Journal of Psychopathology and Behavioral Assessment. 2007;29(3):177-190
- [Background] Brown KW, Ryan RM. The benefits of being present: mindfulness and its role in psychological well-being. J Pers Soc Psychol. 2003 Apr;84(4):822-48. doi: 10.1037/0022-3514.84.4.822. PMID 12703651
- [Background] Buchheld N, Walach H. Mindfulness in Vipassana meditation and psychotherapy - Development of a mindfulness questionnaire. Z Klin Psychol Psych. 2002;50(2):153-172
- [Background] Baer RA, Smith GT, Hopkins J, Krietemeyer J, Toney L. Using self-report assessment methods to explore facets of mindfulness. Assessment. 2006 Mar;13(1):27-45. doi: 10.1177/1073191105283504. PMID 16443717
- [Background] Lai JS, Cella D, Choi S, Junghaenel DU, Christodoulou C, Gershon R, Stone A. How item banks and their application can influence measurement practice in rehabilitation medicine: a PROMIS fatigue item bank example. Arch Phys Med Rehabil. 2011 Oct;92(10 Suppl):S20-7. doi: 10.1016/j.apmr.2010.08.033. PMID 21958919
- [Background] Oude Voshaar MA, ten Klooster PM, Glas CA, Vonkeman HE, Taal E, Krishnan E, Moens HJ, Boers M, Terwee CB, van Riel PL, van de Laar MA. Calibration of the PROMIS physical function item bank in Dutch patients with rheumatoid arthritis. PLoS One. 2014 Mar 17;9(3):e92367. doi: 10.1371/journal.pone.0092367. eCollection 2014. PMID 24637885
- [Background] Condon DM, Revelle W. The international cognitive ability resource: Development and initial validation of a public-domain measure. Intelligence. 2014;43:52-64
- [Background] Holman R, Lindeboom, R., Glas, C. A., Vermeulen, M., & de Haan, R. J. . Constructing an item bank using item response theory: the AMC Linear Disability Score project. Health Services and Outcomes Research Methodology. 2003;4(1):19-33
- [Background] Wainer H. Comparing the incomparable: An essay on the importance of big assumptions and scant evidence. . Educational Measurement: Issues and Practice. 1999;18(4):10-16
- [Background] Reeve BB, Hays RD, Bjorner JB, Cook KF, Crane PK, Teresi JA, Thissen D, Revicki DA, Weiss DJ, Hambleton RK, Liu H, Gershon R, Reise SP, Lai JS, Cella D; PROMIS Cooperative Group. Psychometric evaluation and calibration of health-related quality of life item banks: plans for the Patient-Reported Outcomes Measurement Information System (PROMIS). Med Care. 2007 May;45(5 Suppl 1):S22-31. doi: 10.1097/01.mlr.0000250483.85507.04. PMID 17443115
- [Background] Hansen M, Cai L, Stucky BD, Tucker JS, Shadel WG, Edelen MO. Methodology for developing and evaluating the PROMIS smoking item banks. Nicotine Tob Res. 2014 Sep;16 Suppl 3(Suppl 3):S175-89. doi: 10.1093/ntr/ntt123. Epub 2013 Aug 13. PMID 23943843
- [Background] Hambleton RK, Han N. Assessing the fit of IRT models: Statistical approaches, and the consequences of model misfit. 4/2004, 2004
- [Background] Glas CAW, Suarez-Falcon JC. A comparison of item-fit statistics for the three parameter logistic model. Applied Psychological Measurement. 2003;27:87-107
- [Background] Ponocny I. Nonparametric goodness-of-fit tests for the Rasch model. Psychometrika. 2000;66:437-460
- [Background] Rost J. Rasch models in latent classes: An integration of two approaches to item analysis. Applied Psychological Measurement. 2004;3:271-282
- [Background] Zenisky AL, Hambleton RK, Sireci SG. Identification and evaluation of local item dependencies in the Medical College Admissions Test. Journal of Educational Measurement. 2002;39(4):291-230
- [Background] Samejima F. The graded response model. In: van der Liden WJ, Hambleton R, eds. Handbook of modern item response theory. New York, New York: Springer; 1996:85-100
- [Background] Drasgow F, Levine MV, Tsien S, Williams B, Mead AD. Fitting polytomous item reponse theory models to multiple-choice tests. Applied Psychological Measurement. 1995;19:143-165
- [Background] Choi SW. Firestar: Computerized adaptive testing simulation program for polytomous item response theory models. Appl. Psychol. Meas. 2009;33(8):644
- [Background] Choi SW, Reise SP, Pilkonis PA, Hays RD, Cella D. Efficiency of static and computer adaptive short forms compared to full-length measures of depressive symptoms. Qual Life Res. 2010 Feb;19(1):125-36. doi: 10.1007/s11136-009-9560-5. Epub 2009 Nov 26. PMID 19941077
- [Background] Gershon RC, Rothrock N, Hanrahan R, Bass M, Cella D. The use of PROMIS and assessment center to deliver patient-reported outcome measures in clinical research. J Appl Meas. 2010;11(3):304-14. PMID 20847477
- [Background] Choi SW, Swartz RJ. Comparison of CAT Item Selection Criteria for Polytomous Items. Appl Psychol Meas. 2009 Sep 1;33(6):419-440. doi: 10.1177/0146621608327801. PMID 20011456
- [Background] Kolen MJ, Brennan RL. Test equating, scaling, and linking. Springer; 2004
- [Background] Kim S. A comparative study of IRT fixed parameter calibration methods. Journal of Educational Measurement. 2006;43(4):355-381
- [Background] Thissen D, Varni JW, Stucky BD, Liu Y, Irwin DE, Dewalt DA. Using the PedsQL 3.0 asthma module to obtain scores comparable with those of the PROMIS pediatric asthma impact scale (PAIS). Qual Life Res. 2011 Nov;20(9):1497-505. doi: 10.1007/s11136-011-9874-y. Epub 2011 Mar 8. PMID 21384264
- [Background] Reeve BB, Thissen D, DeWalt DA, Huang IC, Liu Y, Magnus B, Quinn H, Gross HE, Kisala PA, Ni P, Haley S, Mulcahey MJ, Charlifue S, Hanks RA, Slavin M, Jette A, Tulsky DS. Linkage between the PROMIS(R) pediatric and adult emotional distress measures. Qual Life Res. 2016 Apr;25(4):823-33. doi: 10.1007/s11136-015-1143-z. Epub 2015 Sep 30. PMID 26424169
- [Background] Hayes AM, Feldman G. Clarifying the construct of mindfulness in the context of emotion regulation and the process of change in therapy. Clin Psychol-Sci Pr. 2004;11(3):255-262
- [Background] Karam F, Berard A. Reliability and Convergent Validity of the Perceived Stress Scales 4 and 10 Items: Results from the Antidepressants in Pregnancy Discontinuation Study. Pharmacoepidemiology and drug safety. 2009;18:S65-S66
- [Background] Neff KD. The development and validation of a scale to measure self-compassion. Self Identity. 2003;2:223-250
- [Background] Pilkonis PA, Choi SW, Reise SP, Stover AM, Riley WT, Cella D; PROMIS Cooperative Group. Item banks for measuring emotional distress from the Patient-Reported Outcomes Measurement Information System (PROMIS(R)): depression, anxiety, and anger. Assessment. 2011 Sep;18(3):263-83. doi: 10.1177/1073191111411667. Epub 2011 Jun 21. PMID 21697139
- [Background] Guy W. Clinical Global Impressions:ECDEU Assessment Manual for Psychopharmacology. Rockville, MD: National Institute of Mental Health; 1976:218-222
- [Background] Wu PC. Response Shifts in Depression Intervention for Early Adolescents. J Clin Psychol. 2016 Jul;72(7):663-75. doi: 10.1002/jclp.22291. Epub 2016 Mar 18. PMID 26991402
- [Background] Fokkema M, Smits N, Kelderman H, Cuijpers P. Response shifts in mental health interventions: an illustration of longitudinal measurement invariance. Psychol Assess. 2013 Jun;25(2):520-31. doi: 10.1037/a0031669. Epub 2013 Jan 21. PMID 23339313
- [Background] Oort FJ. Using structural equation modeling to detect response shifts and true change. Qual Life Res. 2005 Apr;14(3):587-98. doi: 10.1007/s11136-004-0830-y. PMID 16022054
- [Background] Nolte S, Elsworth GR, Sinclair AJ, Osborne RH. Tests of measurement invariance failed to support the application of the "then-test". J Clin Epidemiol. 2009 Nov;62(11):1173-80. doi: 10.1016/j.jclinepi.2009.01.021. Epub 2009 Jul 12. PMID 19595570
- [Background] Barclay-Goddard R, Lix LM, Tate R, Weinberg L, Mayo NE. Response shift was identified over multiple occasions with a structural equation modeling framework. J Clin Epidemiol. 2009 Nov;62(11):1181-8. doi: 10.1016/j.jclinepi.2009.03.014. Epub 2009 Jul 16. PMID 19615858
- [Background] Schwarz N, Oyserman D. Asking questions about behavior: Cognition, communication, and questionnaire construction. Am J Eval. 2001;22(2):127-160
- [Background] Guyatt GH, Osoba D, Wu AW, Wyrwich KW, Norman GR; Clinical Significance Consensus Meeting Group. Methods to explain the clinical significance of health status measures. Mayo Clin Proc. 2002 Apr;77(4):371-83. doi: 10.4065/77.4.371. PMID 11936935
- [Background] Hays RD, Woolley JM. The concept of clinically meaningful difference in health-related quality-of-life research. How meaningful is it? Pharmacoeconomics. 2000 Nov;18(5):419-23. doi: 10.2165/00019053-200018050-00001. PMID 11151395
- [Background] Norman GR, Sridhar FG, Guyatt GH, Walter SD. Relation of distribution- and anchor-based approaches in interpretation of changes in health-related quality of life. Med Care. 2001 Oct;39(10):1039-47. doi: 10.1097/00005650-200110000-00002. PMID 11567167
- [Background] Crosby RD, Kolotkin RL, Williams GR. Defining clinically meaningful change in health-related quality of life. J Clin Epidemiol. 2003 May;56(5):395-407. doi: 10.1016/s0895-4356(03)00044-1. PMID 12812812
- [Background] Hays RD, Revicki DA. Reliability and Validity (including Responsiveness). In: Fayers P, Hays RD, eds. Quality of Life Assessment in Clinical Trials. 2nd ed. Oxford: Oxford University Press; 2005:25-40
- [Background] Sloan JA, Cella D, Hays RD. Clinical significance of patient-reported questionnaire data: another step toward consensus. J Clin Epidemiol. 2005 Dec;58(12):1217-9. doi: 10.1016/j.jclinepi.2005.07.009. Epub 2005 Oct 13. No abstract available. PMID 16291464
- [Background] MacCallum RC, Widaman KF, Preacher KJ, Hong S. Sample Size in Factor Analysis: The Role of Model Error. Multivariate Behav Res. 2001 Oct 1;36(4):611-37. doi: 10.1207/S15327906MBR3604_06. PMID 26822184
- [Background] Wolf EJ, Harrington KM, Clark SL, Miller MW. Sample Size Requirements for Structural Equation Models: An Evaluation of Power, Bias, and Solution Propriety. Educ Psychol Meas. 2013 Dec;76(6):913-934. doi: 10.1177/0013164413495237. PMID 25705052
- [Background] Bentler PM, Chou C-P. Practical issues in structural modeling. Sociological Methods & Research. 1987;16(1):78-117
- [Background] Nunnally JC, Bernstein IH, Berge JMt. Psychometric theory. Vol 226: JSTOR; 1967
- [Background] Hays RD, Revicki D, Coyne KS. Application of structural equation modeling to health outcomes research. Eval Health Prof. 2005 Sep;28(3):295-309. doi: 10.1177/0163278705278277. PMID 16123259
- [Background] Schwartz CE, Ahmed S, Sawatzky R, Sajobi T, Mayo N, Finkelstein J, Lix L, Verdam MG, Oort FJ, Sprangers MA. Guidelines for secondary analysis in search of response shift. Qual Life Res. 2013 Dec;22(10):2663-73. doi: 10.1007/s11136-013-0402-0. Epub 2013 Apr 10. PMID 23572398
- [Background] Schwartz CE, Sprangers MA, Oort FJ, Ahmed S, Bode R, Li Y, Vollmer T. Response shift in patients with multiple sclerosis: an application of three statistical techniques. Qual Life Res. 2011 Dec;20(10):1561-72. doi: 10.1007/s11136-011-0056-8. Epub 2011 Nov 13. PMID 22081216
- [Background] King-Kallimanis BL, Oort FJ, Visser MR, Sprangers MA. Structural equation modeling of health-related quality-of-life data illustrates the measurement and conceptual perspectives on response shift. J Clin Epidemiol. 2009 Nov;62(11):1157-64. doi: 10.1016/j.jclinepi.2009.04.004. PMID 19595574
- [Background] Visser MR, Oort FJ, Sprangers MA. Methods to detect response shift in quality of life data: a convergent validity study. Qual Life Res. 2005 Apr;14(3):629-39. doi: 10.1007/s11136-004-2577-x. PMID 16022057
- [Background] Cella DF, Gonin R, Lloyd S. The Q-SCORE: Scaling the Tower of Babel in Quality of Life (QL) Measurement